CLINICAL TRIAL: NCT06885840
Title: A Multi-cohort, Open-label Phase II Study to Evaluate the Efficacy and Safety of the Anti-EGFR/c-Met Bispecific Antibody MCLA-129 in Patients with Advanced Non-Small Cell Lung Cancer with Actionable Gene Alterations and MET Amplification.
Brief Title: Study of MCLA-129 in the Treatment of Advanced Non-small Cell Lung Cancer with AGA and MET Amplification.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTP-21723
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): Patients with advanced NSCLC with previously detected EGFR-sensitive mutations (exon 19 deletion or exon 21 L858R mutation) who have progressed after prior standard treatment and with MET amplification after failure of treatment with EGFR-TKIs.
  Interventions: Drug: MCLA-129
- Cohort 2 (Experimental): Patients with advanced NSCLC with previously detected EGFR-sensitive mutations (exon 19 deletion or exon 21 L858R mutation) who have progressed after prior standard treatment and with disease progression or intolerance after MET inhibitors and who have benefited from such treatment.
  Interventions: Drug: MCLA-129
- Cohort 3 (Experimental): Patients with advanced NSCLC with previously detected actionable gene alterations who had progressed after treatment with corresponding inhibitors and platinum-based chemotherapy also with MET amplification after failure of treatment with the corresponding driver gene inhibitors.
  Interventions: Drug: MCLA-129
- Cohort 4 (Experimental): Patients with advanced NSCLC with previously detected actionable gene alterations who had progressed after treatment with corresponding inhibitors, platinum-based chemotherapy and with disease progression or intolerance after MET inhibitors and who have benefited from such treatment.
  Interventions: Drug: MCLA-129

INTERVENTIONS:
Drug: MCLA-129 — MCLA-129 will be administered by intravenous infusion on the 28-day treatment cycle.

SUMMARY:
This is a multi-center, open-label, phase II clinical study of MCLA-129 as monotherapy in patients with advanced non-small cell lung cancer (NSCLC) with actionable gene alterations and MET amplification to evaluate the efficacy, safety, pharmacokinetic characteristics of MCLA-129.

DETAILED DESCRIPTION:
This is a multi-center, open-label, monotherapy, multi-cohort phase II study of MCLA-129 in patients with advanced non-small cell lung cancer (NSCLC) with actionable gene alterations and MET amplification, designed to evaluate the efficacy, safety, and PK profiles of MCLA-129 in the target population.

Subjects who must experience disease progression or intolerance after standard treatment eligible through screening will be divided into the following 4 cohorts:

Cohort 1 and Cohort 2: Patients with advanced NSCLC with previously detected EGFR-sensitive mutations (exon 19 deletion or exon 21 L858R mutation) who have progressed after prior standard treatment which includes 1) first-generation or second-generation EGFR-TKIs, with T790M mutation requiring third-generation EGFR-TKIs and platinum-based chemotherapy; or 2) first-generation or second-generation EGFR-TKIs, with T790M mutation negative or unknown status.

Subjects in Cohort 1: Patients with MET amplification after failure of treatment with EGFR-TKIs.

Subjects in Cohort 2: Patients who experienced disease progression or intolerance after MET inhibitors and benefited from such treatment.

Cohort 3 and Cohort 4: Patients with advanced NSCLC with previously detected actionable gene alterations who had progressed after treatment with corresponding inhibitors and platinum-based chemotherapy.

Subjects in Cohort 3: Patients with MET amplification, after failure of treatment with the corresponding driver gene inhibitors.

Subjects in Cohort 4 should also meet: Patients who experienced disease progression or intolerance after MET inhibitors and benefited from such treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are ≥ 18 years of age, regardless of gender.
* Subjects must have histologically or cytologically confirmed locally advanced unresectable or metastatic NSCLC.
* Subjects who must experience disease progression or intolerance after standard treatment eligible through screening will be divided into the following 4 cohorts:

Cohort 1 and Cohort 2: Patients with advanced NSCLC with previously detected EGFR-sensitive mutations (exon 19 deletion or exon 21 L858R mutation) who have progressed after prior standard treatment which includes 1) first-generation or second-generation EGFR-TKIs, with T790M mutation requiring third-generation EGFR-TKIs and platinum-based chemotherapy; or 2) first-generation or second-generation EGFR-TKIs, with T790M mutation negative or unknown status.

Subjects in Cohort 1: Patients with MET amplification after failure of treatment with EGFR-TKIs.

Subjects in Cohort 2: Patients who experienced disease progression or intolerance after MET inhibitors and benefited from such treatment.

Cohort 3 and Cohort 4: Patients with advanced NSCLC with previously detected actionable gene alterations who had progressed after treatment with corresponding inhibitors and platinum-based chemotherapy.

Subjects in Cohort 3: Patients with MET amplification after failure of treatment with the corresponding driver gene inhibitors.

Subjects in Cohort 4: Patients who experienced disease progression or intolerance after MET inhibitors and benefited from such treatment.

* Subjects must have measurable lesions that meet the definition of RECIST v1.1. Selected target lesions must meet one of the following two criteria: 1) no prior local therapy or radiation or 2) subsequent progression occurs within the prior local therapy area as determined by RECIST v1.1..
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Expected survival ≥3 months.
* Have certain functions of organ systems (no blood transfusion or use of blood component or G-CSF support within 14 days before testing), defined as follows:

  * Absolute neutrophil count (ANC) ≥1.5×10^9 /L.
  * Platelet count (PLT）≥75×10^9 /L.
  * Hemoglobin (HGB) ≥100 g/L.
  * Serum albumin ≥ 30 g/L.
  * Total bilirubin ≤1.5 times the upper limit of normal (ULN).
  * Alanine amino transferase (ALT) and aspartate amino transferase (AST) ≤3×ULN.
  * Creatinine ≤1.5×ULN. If creatinine is >1.5×ULN, creatinine clearance ≥50 mL/min as calculated by Cockcroft-Gault formula, or 24-hour urine creatinine clearance ≥50 mL/min is measured, the patients can still be enrolled.
* Willing and able to follow the trial and follow-up procedures.
* Able to understand the nature of the trial and voluntarily sign the written informed consent form.

Exclusion Criteria:

* Have received an investigational product or antitumor drug treatment (including known anti-tumor traditional Chinese medicine treatment) within 14 days before the first dose of MCLA-129 or within 5 half-lives of the drug (whichever is longer) (for a drug with a long half-life, it is required that the interval from the last dose to be at most 4 weeks; for chemotherapy with delayed toxicity, such as nitrosourea or mitomycin C, it shall be 6 weeks before [the treatment]).
* Have undergone a major surgery and radiotherapy (local palliative radiotherapy is allowed 2 weeks or more prior to the first dose) within 4 weeks prior to the first dose of MCLA-129.
* Have previously received systemic anti-tumor therapy beyond the fourth line (excluding maintenance therapy).
* Prior use of EGFR/c-Met bispecific antibody or ADC drugs (Amivantamab [JNJ-61186372], EMB-01, GB263T, PM1080/HS-20117, TAVO412, YH013/DM005, AZD9592, or SHR-9839).
* Prior to the first dose of MCLA-129, previous treatment-related toxicities have not resolved to Grade 1 or below (CTCAE 5.0 criteria), except for alopecia.
* Prior to the first dose of MCLA-129, previous treatment-related toxicities have not resolved to Grade 1 or below (CTCAE 5.0 criteria), except for alopecia.
* Have had other malignancies within the past 3 years, except for cancers that have been totally cured or locally cured, such as basal or squamous cell carcinoma of the skin, cervical cancer in situ, or breast cancer in situ.
* Patients with primary malignant tumor of central nervous system, or metastases to meninges, or concomitantly with symptomatic brain metastases, or new therapy naive brain metastases.

Note: Patients with brain metastases who have received treatment for brain metastases (including systemic and local therapies against brain metastases) with no obvious symptoms and stable condition, and do not require drug therapy such as steroids and/or dehydration to reduce intracranial pressure within 2 weeks before enrollment and have no risk of brain bleeding can be enrolled.

* With clinically significant cardiovascular and cerebrovascular diseases.

  * Arterial thromboembolism, deep vein thrombosis or lung embolism diagnosed within 3 month before first administration of the investigational drug. Non-obstructive catheter related clot and other clinically irrelevant thrombosis are not included in the exclusion criteria. Patients with a history of related thrombosis diagnosed 3 months ago must be clinically stable for at least 4 weeks before initial administration.
  * With any of the following medical history within 6 months before first administration of the investigational drug: myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary or peripheral artery bypass, or any acute coronary syndrome.
  * With abnormal ECG corrected QT interval (QTcF) at rest in the screening period. Remeasurement is made twice at intervals of more than 5 minutes. For average QTcF of 3 ECG inspections: male: ≥ 450 msec, and female: ≥ 470 msec. With clinically significant abnormal heart rate, conduction, and ECG form at rest, e.g. complete left bundle branch block, third-degree conduction block, second-degree conduction block, and PR interval > 250 msec, double law, triple law, preexcitation syndrome, etc.
  * Poorly controlled hypertension in the investigator's opinion (systolic blood pressure > 180 mmHg, or diastolic blood pressure > 100 mmHg).
  * New York Heart Association Grade III-IV congestive heart failure, or hospitalization due to congestive heart failure within 6 months before first administration of the investigational drug.
  * Pericarditis/clinically significant pericardial effusion.
  * Cardiomyopathy.
  * Other clinically significant cardiovascular disorders as believed by investigators.
* Active hepatitis B (positive hepatitis B surface antigen (HBsAg) and serum HBV DNA ≥ 2,000 IU/mL [equivalent to 104 copies/mL]), positive hepatitis C virus antibody, HIV antibody and treponema pallidum antibody.
* Subjects with a history of interstitial lung disease or current clinical evidence of interstitial lung disease, including drug-induced Interstitial lung disease or radiation pneumonitis.
* Presence of a serious disease or medical condition currently, including but not limited to uncontrolled active infection, uncontrolled pleural or peritoneal effusion, and clinically significant pulmonary, metabolic or psychiatric diseases.
* Females of childbearing potential, pregnant or breastfeeding women with a positive serum pregnancy test 7 days before the start of treatment, and male and female subjects who are unwilling to use effective contraceptive measures or plan to have a child throughout the treatment period and within 3 months after the end of treatment.
* Patients with known allergic reactions and hypersensitivity reactions, or be allergic to MCLA-129 or any of its excipients.
* Patients with poor compliance, inability or unwillingness to follow the study and/or follow-up procedure listed in the protocol, or patients who are not suitable to participate in this trial, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 at RP2D in patients with advanced NSCLC and other solid tumors in each cohort in Part 2 in terms of overall response rate (ORR)

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years.
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of clinical benefit rate (CBR).
Disease Control Rate (DCR) | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years.
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of disease control rate (DCR)
Progression-Free Survival (PFS) | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years.
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of progression-free survival (PFS).
Duration of Response (DOR) | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years.
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of duration of response (DOR).
Time to response (TTR) | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years.
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of time to response (TTR).
Overall Survival (OS) | From date of first treatment every 6 weeks until death or withdrawal, whichever came first, approximately 2 years.
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of overall survival (OS).
Treatment-Emergent Adverse Event (TEAE) | Until 30 days after the last dosing
  To evaluate the safety of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of treatment-emergent adverse event (TEAE).
Area under the concentration versus time curve [AUC0-∞] | : Until 30 days after the last dosing.
  To evaluate the population PK profile of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of area under the concentration versus time curve [AUC0-∞].
Anti-Drug Antibody (ADA) | Until 30 days after the last dosing.
  To assess the Incidence of anti-drug antibodies in serum blood against MCLA-129 following administration of MCLA-129.

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Foshan First People's Hospital, Foshan, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Hebei University Affiliated Hospital, Baoding, Hebei
  - Harbin Medical University Affiliated Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nantong Cancer Hospital, Nantong, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Chest Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No